CLINICAL TRIAL: NCT04611984
Title: Osteocalcin and Cross-Linked C-Terminal Telopeptides of Type I Collagen in Gingival Crevicular Fluid During Piezocision Accelerated Orthodontic Tooth Movement
Brief Title: OC and ICTP in Gingival Crevicular Fluid During Piezocision Accelerated Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 04.03.2013.38
Record Dates: First submitted 2020-10-20; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Tooth Movement
Keywords: Tooth movement; Piezocision; Gingival crevicular fluid; Osteocalcin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators performing the clinical and surgical procedures, and patients were not blinded. Data assessment was performed by a blinded researcher. Gingival crevicular fluid samples were collected and numbered by another blinded researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezocision (Experimental): Piezocision was performed on the mesial and distal side of the maxillary right canine tooth which was served as the piezocision group. Then canine distalization was performed via closed-coil springs applying 150 g of force by using mini-screws as anchorage.
  Interventions: Procedure: Piezocision
- Control (Active Comparator): Maxillary left canine served as the control group and canine distalization was performed via closed-coil springs applying 150 g of force by using mini-screws as anchorage.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Piezocision — Piezocisions were performed on the mesial and distal sides of the right maxillary canines. Then canine distalization was performed via closed-coil springs applying 150 g of force by using mini-screws as anchorage.
  Arms: Piezocision
Procedure: Control — The mesial and distal sides of the left maxillary canines served as controls and canine distalization was performed via closed-coil springs applying 150 g of force by using mini-screws as anchorage.
  Arms: Control

SUMMARY:
The aim of this study was to evaluate the tooth movement with and without piezocision with regard to the levels of osteocalcin and cross-linked C-terminal telopeptides of type I collagen in the gingival crevicular fluid.

DETAILED DESCRIPTION:
15 systemically healthy subjects requiring extraction of the maxillary 1. premolars with distalization of the maxillary canines were enrolled to the study. Piezocisions were performed on the distal and mesial sides of the right maxillary canines while the left maxillary canines served as controls. Canine distalization was performed via closed-coil springs applying 150 g of force per side by using miniscrews as anchorage. Gingival crevicular fluid samples were collected from both mesial and distal sides of right and left maxillary canines at 0, 1, 7, 14 and 28 days. The gingival crevicular fluid levels of osteocalcin and cross-linked C-terminal telopeptides of type I collagen were determined by using ELISA. The rate of tooth movement was measured on 14 and 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Class I, Class II or Class III malocclusion,
* Proclined incisors requiring extraction of the maxillary first premolars with subsequent retraction of the maxillary canines
* No previous orthodontic treatment
* Good oral hygiene and periodontal health (plaque and gingival indices less or equal 1, probing depth less or equal 3 mm, no radiographic bone loss).

Exclusion Criteria:

* having systemic diseases that could affect bone and tooth movement
* smoking

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid osteocalcin level (ng/ml) | 28 days after canine distalization
  Gingival crevicular fluid samples were collected from mesial and distal sides of the maxillary right and left canines.The gingival crevicular fluid level of osteocalcin was determined by using ELISA
Gingival crevicular fluid cross-linked C-terminal telopeptides of type I level (ng/ml) | 28 days after canine distalization
  Gingival crevicular fluid samples were collected from mesial and distal sides of the maxillary right and left canines.The gingival crevicular fluid level of cross-linked C-terminal telopeptides of type I collagen was determined by using ELISA.

SECONDARY OUTCOMES:
The amount of canine movement (mm) | Baseline (day 0) before canine distalization and, 14 and 28 days after canine distalization
  All measurements were performed on the dental cast model using a digital caliper. The amount of space closure was based on the measurements of the distance between the contact points of the distal surface of canine and the mesial surface of second premolar. The change of distance between the three observation periods represented the amount of canine movement.
Retraction rate (mm/day) of canine movement | 14 and 28 days after canine distalization
  All measurements were performed on the dental cast model using a digital caliper. The amount of space closure was based on the measurements of the distance between the contact points of the distal surface of canine and the mesial surface of second premolar. The change of distance between the three observation periods represented the amount of canine movement, which was divided by the number of days between two sessions to obtain the retraction rate on daily basis

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Selin Yıldırım, Dr., Principal Investigator — Marmara University, Faculty of Dentistry, Department of Peridontology
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Dibart S, Surmenian J, Sebaoun JD, Montesani L. Rapid treatment of Class II malocclusion with piezocision: two case reports. Int J Periodontics Restorative Dent. 2010 Oct;30(5):487-93. PMID 20814602
- [Background] Alfaqeeh SA, Anil S. Osteocalcin and N-telopeptides of type I collagen marker levels in gingival crevicular fluid during different stages of orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2011 Jun;139(6):e553-9. doi: 10.1016/j.ajodo.2011.03.005. PMID 21640867
- [Background] Raj SC, Praharaj K, Barik AK, Patnaik K, Mahapatra A, Mohanty D, Katti N, Mishra D, Panda SM. Retraction With and Without Piezocision-Facilitated Orthodontics: A Randomized Controlled Trial. Int J Periodontics Restorative Dent. 2020 Jan/Feb;40(1):e19-e26. doi: 10.11607/prd.3968. PMID 31815981